CLINICAL TRIAL: NCT01916603
Title: Effectiveness of a Normative Intervention (Diet, Physical Activity and Breastfeeding) on Maternal Nutrition and Offspring Growth and Development: Nutrition in the First 1000 Days Key to Healthy Growth and Long-term Health.
Brief Title: Diet, Physical Activity and Breastfeeding Intervention on Maternal Nutrition, Offspring Growth and Development
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Chile (Other)
Collaborators: National Nutrition and Food Technology Institute (Other); Pontificia Universidad Catolica de Chile (Other); Fondo Nacional de Desarrollo Científico y Tecnológico, Chile (Other Government); Ministry of Health, Chile (Other Government)
Responsible Party: Principal Investigator, Ricardo Uauy, Ph.D. Doctor in Philosophy, University of Chile
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: Fondecyt #1130277
Record Dates: First submitted 2013-07-04; First posted 2013-08-05 (Estimated); Last update posted 2013-08-05 (Estimated); Status verified 2013-07

CONDITIONS: Obesity; Weight Gain; Metabolic Diseases; Birth Weight; Infant Nutrition Disorders
MeSH Terms: conditions — Obesity; Weight Gain; Metabolic Diseases; Birth Weight; Infant Nutrition Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Normative intervention (Experimental): Normative intervention on diet & physical & breastfeeding: diet and physical activity counselling-support and breastfeeding promotion till 12 months postpartum
  Interventions: Behavioral: Normative Intervention
- Routine care (No Intervention): Routine antenatal care according to national guidelines

INTERVENTIONS:
Behavioral: Normative Intervention — Diet and physical activity counselling-support and breastfeeding promotion till 12 months postpartum
  Arms: Normative intervention

SUMMARY:
NCDs are observed mostly in adults, however there is strong evidence that suggests NCDs origin early in life, thus the first 1000 days of life (conception to age 2yrs). Studies show that maternal BMI before conception and during pregnancy predict future risk of obesity and associated metabolic conditions in both mother and offspring. Weight gain during the first two years of life is also critical in defining the infant's predisposition to obesity during adulthood. Objective: to assess the effectiveness of delivering a primary health care intervention to enhance compliance with updated nutrition and health care (diet, physical activity and breastfeeding) standards from early pregnancy through the first year of life. Methods: cluster randomized controlled trial (CRCT), designed as a public health intervention "program effectiveness" study (i.e. intervention will be available through the established national health system under standard operating conditions). A cluster unit will be a primary health care centers (PHCC) in South-East Santiago 12 PHCC will be randomly allocated to: enhanced nutrition and health care (intervention group) or routine nutrition and health care (control group).We will recruit 200 women in each of 12 PHCC; assuming a 20% loss to f-up we will complete 960 women per arm. After randomization, pregnant women in the intervention PHCCs starting at their first pre-natal visit (< 15 wks.) will receive, diet and physical activity (PA) counseling-support based on updated recommendations and monitoring goals for weight gain & glycemic control and breastfeeding (BF) promotion till 12 m postpartum. Pregnant women who attend control PHCCs will receive routine antenatal care according to national guidelines. Expected results: participants in the intervention PHCCs will benefit by achieving adequate nutritional status & metabolic control, during and early after, pregnancy as well as adequate infant growth & development as a result of improved nutrition and health care practices. The results will likely be generalizable through the primary health care system; considering this is a "program effectiveness" trial conducted under "real life" conditions . Additionally, we will include specific ancillary mechanistic projects to better characterize the intervention and its impact.

DETAILED DESCRIPTION:
Introduction: in Chile as well as in most of the world, obesity and related chronic diseases (cardiovascular diseases, cancer and diabetes (NCDs)) are presently the main causes of death and disability. Although these conditions are observed mostly in adulthood, there is now considerable evidence that indicates that they are rooted in the first 1000 days of life (from -1 to + 2yrs of life).

Several studies show that maternal BMI before conception and during pregnancy predict future risk of obesity and associated metabolic conditions for both mother and offspring. Weight gain during the first two years of life is also critical, not only to ensure infant survival, but also in defining the infant's predisposition to the emergence of chronic diseases during adulthood. From a population perspective, the most effective approach to counteract the epidemic of obesity and NCDs is to prevent them. Recommendations for healthy diets and physical activity during pregnancy and infancy, as well as monitoring of nutrition goals are currently available in the Chilean primary health care system. However, most of these recommendations are not up to date and virtually all are poorly implemented. Objective: to assess the effectiveness of delivering (via primary health centers) an intervention that enhances compliance with up to date nutrition and health care standards (regarding diet, physical activity and breastfeeding promotion) during pregnancy and the first year of life. The main goal is that mothers achieve adequate nutritional status & metabolic control, during and early after pregnancy, and that infants grow and develop healthily (adequate linear and ponderal growth according to WHO standard, while avoiding excess BMI gains) Methods: this is a cluster randomized controlled trial (CRCT), designed as a public health "program effectiveness" study (i.e. intervention will be available through the established national health system under standard operating conditions). The cluster units will be 12 primary health care centers (PHCC) in South-East Santiago randomly allocated to: 1) enhanced nutrition and health care standards (intervention group) or 2) routine care (control group).

Women seeking care before 15 weeks of pregnancy, residents within a catchment area of selected PHCCs, who are not planning to move in the next two years will be invited to participate in the study. Pregnant women classified as high risk according to the norms of the Chilean Ministry of Health (MoH)and/or underweight (BMI<18.5) will be excluded. We will recruit 200 women in each PHCC and assuming a 20% loss to f-up we will end with 960 women per arm of the study. After randomization, pregnant women in the intervention PHCCs starting at their first pre-natal visit (< 15 wks.) will receive, diet and physical activity (PA) counseling-support based on updated recommendations and monitoring goals for weight gain & glycemic control and breastfeeding (BF) promotion till 12 months postpartum. Pregnant women who attend control PHCCs will receive routine antenatal care according to national guidelines. The outcomes will be: 1)achievement of adequate nutritional status & metabolic control during pregnancy: a. Weight gain according to Institute of Medicine (IOM) recommendations, b. glycemic control based on ADA 2011 recommendations, 3. No weight retention at 12 months, and 2) healthy infant growth and development: a) height and BMI growth based on WHO standards, b) normal abbreviated psychomotor development test (TEPSI) and evaluation scale of psychomotor development (EEDP) at 12 months. Mothers & infants will be monitored to ensure the safety of the intervention (assessment of undernutrition, micronutrient deficiency and indices of poor nutrition). Data will be collected as part of routine health care activities and analyzed based on the allocation to each study group ("intention to treat"). Results will be presented as appropriate effect sizes with a measure of precision (95% confidence intervals). Further exploratory analyses will be based on those participants that fully follow the protocol ("per-protocol analyses"). Expected results: we expect that the intervention will benefit the participants in achieving adequate nutritional status & metabolic control, during and early after, pregnancy as well as adequate infant growth & development as a result of an increase in the impact of standard nutrition and health care practices. The results should be potentially extended to the rest of the primary health care system given the "program effectiveness" approach that will be taken. Additionally, we expect that this study will serve as a core project in which other ancillary projects will be nested. Gathered information should contribute to a better understanding of how to develop effective interventions to halt the maternal and obesity epidemic and its associated co-morbidities in the Chilean population.

ELIGIBILITY:
Inclusion Criteria:

* Women seeking care before 15 weeks of pregnancy, residents within catchment area of selected Primary Health Care Centers, who are not planning to move in the next two years will be invited to participate in the study

Exclusion Criteria:

* Pregnant women classified as high risk according to the norms of the Chilean Ministry of Health(MoH) and/or underweight (BMI<18.5)

Ages: 16 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2400 (Estimated)
Dates: Start 2013-09; Primary Completion 2013-09 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Weight gain and nutritional status in mothers | 36-40 weeks of gestation
Weight retention | 12 months post-partum
Glycaemic control | At 20-24 weeks of pregnancy
Lactation rates | At 12 months post-partum
Initiation and duration of breastfeeding (exclusive and total) | Birth-12 months
Weight, length and BMI growth in infants | During the first year of life
Psychomotor development (based on abbreviated scale) | During the first year of life

SECONDARY OUTCOMES:
Implementation | At 30 months into the recruitment
  Implementation: compliance to protocol by health personnel, midwives & dieticians per center, time allocated to the actions of the interventions, etc.
Participant compliance variables | At 30 months into the recruitment
  Variables relate to the adoption by participants of the respective program activities: adherence to diet/physical activity prescriptions, adequate referral, attendance to dietician's clinic, lactation workshops, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Uauy, PhD, Principal Investigator — University of Chile
Locations (1):
- Institute of Nutrition and Food Technology, Santiago, Santiago Metropolitan, Chile

REFERENCES:
- [Derived] Mujica-Coopman MF, Corvalan C, Flores M, Garmendia ML. The Chilean Maternal-Infant Cohort Study-II in the COVID-19 Era: A Study Protocol. Front Public Health. 2022 Jul 14;10:904668. doi: 10.3389/fpubh.2022.904668. eCollection 2022. PMID 35910889
- [Derived] Garmendia ML, Corvalan C, Araya M, Casanello P, Kusanovic JP, Uauy R. Effectiveness of a normative nutrition intervention in Chilean pregnant women on maternal and neonatal outcomes: the CHiMINCs study. Am J Clin Nutr. 2020 Oct 1;112(4):991-1001. doi: 10.1093/ajcn/nqaa185. PMID 32692805
- [Derived] Garmendia ML, Mondschein S, Matus O, Murrugarra R, Uauy R. Predictors of gestational weight gain among Chilean pregnant women: The Chilean Maternal and Infant Nutrition Cohort study. Health Care Women Int. 2017 Aug;38(8):892-904. doi: 10.1080/07399332.2017.1332627. Epub 2017 May 19. PMID 28524735
- [Derived] Garmendia ML, Corvalan C, Araya M, Casanello P, Kusanovic JP, Uauy R. Effectiveness of a normative nutrition intervention (diet, physical activity and breastfeeding) on maternal nutrition and offspring growth: the Chilean maternal and infant nutrition cohort study (CHiMINCs). BMC Pregnancy Childbirth. 2015 Aug 18;15:175. doi: 10.1186/s12884-015-0605-1. PMID 26283529